CLINICAL TRIAL: NCT04504981
Title: HIV Prevention for High Risk African American Young Men
Brief Title: Y2Prevent: Preventing Drug Use and HIV Through Empowerment, Social Support and Mentorship (Y2P)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Michele D. Kipke, Profrssor of Pediatrics, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHLA-19-00029; R34DA044106 (NIH)
Record Dates: First submitted 2020-08-03; First posted 2020-08-07 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: HIV; Drug Use

STUDY DESIGN:
Intervention Model Description: In Phase 3, we will pilot test Y2Prevent with three groups of African American young men who have sex with men (AAYMSM) in Los Angeles. Each group will have up to 10 members (n=30). The intervention will be delivered to the three groups in a sequential order so that the experiences from the first group can be used to adapt and/or further refine the intervention before it is pilot tested with the second group. Feedback from the first group will be used to further adapt and refine the intervention. It will be pilot tested again with a second group of 10 participants. Y2Prevent will be further refined as needed, and it will then be pilot tested with a third and final group of up to ten participants.
Masking Description: This is a pilot study with no comparison/control group so masking is not relevant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Y2Prevent Intervention (Other): Y2Prevent will include several intervention components (i.e., My Legacy, Sources of Influence, Healthy Relationships, Goal Setting, Health and Self-Efficacy, and Mentorship). These intervention components are intended to assist participants: a) explore future adult identity and envision a positive future, b) develop behavioral skills related to problem-solving and goal-setting, c) develop behavioral skills related to communication, negotiation and conflict resolution with romantic and sexual partners, d) identify ways to safeguard their future by taking responsibility for their health, e) obtain information about HIV transmission and HIV prevention, including HIV testing, treatment as prevention (TaSP) and the availability of PrEP and PEP for prevention, and f) a participant-identified mentor to provide support and encouragement related to behavior change and implementing their future goals and plans.
  Interventions: Behavioral: Y2Prevent

INTERVENTIONS:
Behavioral: Y2Prevent — Y2Prevent (Y2P) is a groupl level intervention that consists of 7 weekly group sessions focused on helping young African American men who have sex with men (AAYMSM) identify life goals and safeguard their health to achieve those goals

SUMMARY:
The goal of this clinical trial is to pilot test a group level intervention, called Y2Prevent, which aims to decrease drug use and HIV/STI risk among Black/African American young men who have sex with men (AAYMSM). The main question it aims to answer is:

• determine if Y2Prevent is possible to engage in easily and is accepted by the participants, for potential expansion to other cities.

Participants will engage in 7 weekly group sessions focused on helping AAYMSM identify life goals and safeguard their health to achieve those goals. This intervention will also include:

* HIV/STI testing and treatment referral
* drug screening and treatment referral
* positive youth development and future planning through a mentorship program

DETAILED DESCRIPTION:
The overarching aim is to develop a culturally tailored and developmentally appropriate HIV prevention intervention for African American young men who have sex with men (AAYMSM), ages 18 to 24 years. No group is at greater risk for acquiring HIV than YMSM, especially those living in inner cities, with AAYMSM now accounting for the largest number of new HIV infections detected in cities each year. If these trends continue, it is estimated that as many as 1 in 2 AAYMSM will be diagnosed with HIV in their lifetime.

The investigators propose to further refine and pilot test an intervention, called Young Men's Adult Identity Mentoring (YM-AIM). Adapted from an existing CDC Diffusing Effective Behavioral Intervention (DEBI), YM-AIM is a theory-driven, group-level intervention designed to help AAYMSM develop a healthy vision for their future (or "possible future self") by defining a set of short- and long-term goals in the areas of education, health, family and intimate relationships. Through the facilitated activities, participants consider how their involvement in risky behaviors (e.g., illicit drug use, condomless sex, multiple sex partners) would interfere with achieving those goals. With funding from NIDA (R21 DA024588), the investigators developed YM-AIM in response to findings from our own research, as well as those reported in the literature, which demonstrate that experiences of minority stress (e.g., racism, homophobia) and exposure to violence and victimization (family, intimate partner, community) put AAYMSM at significantly greater risk for illicit drug use, HIV/STI sexual risk (condomless anal sex), and mental health problems (e.g., depression) as compared to Caucasian and Hispanic/Latino YMSM.

During our initial pilot, participants (n=36) were enormously enthusiastic about their participation in YM-AIM (all participants attended all six weekly sessions), they provided positive feedback about the various components, activities, and exercises, and they reported that YM-AIM should continue to be delivered using a group-based intervention because they enjoyed the support provided by other group members. Participants also reported they wanted (and needed) ongoing social support after completing the intervention, to help them achieve their short- and long-term goals and maintain positive changes in sexual risk behaviors. This feedback is consistent with the literature that suggests mentors are immensely beneficial, particularly for youth and young adults, because they can share their worldviews, experiences, knowledge, support and advice, as well as provide a positive influence. By introducing youth to new experiences and sharing positive values, mentors can help young people avoid negative behaviors and achieve success. Having a mentor has also been found to reduce youths' risk for delinquency, aggression and drug use and lead to increased academic satisfaction and performance. Based on this, the investigators propose to further strengthen and refine YM-AIM by adding a youth mentoring/support component, called Youth Initiated Mentoring (YIM). YIM uses a positive youth development framework to help young, low-income ethnic/racial minorities: a) build social capital to achieve immediate and long-term life goals, b) build social support networks, c) identify and engage natural mentors in their networks to address structural barriers encountered in their lives, and d) develop relationships with supportive adults.

YM-AIM was developed in 2011, before widespread availability of PrEP/PEP. The investigators are therefore also proposing to add three new components: 1) biomedical HIV prevention strategies (PrEP, PEP), 2) HIV/STI testing and treatment referral, and 3) drug screening and treatment referral. This new intervention, which is called Y2Prevent, will then be evaluated for its feasibility and acceptability. Intervention outcomes include drug use in past 30 days and 3 months, alcohol use, condomless sex, number of partners, condom use intention, condom use self-efficacy, HIV testing recency/frequency, and linkage to care. The specific aims are to:

SPECIFIC AIM 1: Conduct formative research to develop Y2Prevent and refine our assessment measures.

SPECIFIC AIM 2: Finalize Y2Prevent study protocols and consents and develop a manual of operations.

SPECIFIC AIM 3: Pilot and evaluate Y2Prevent to determine intervention feasibility and acceptability, and collect prelimiary efficacy data.

e propose to integrate YM-AIM and YIM into a single new intervention, called Y2Prevent. This intervention will then be implemented and evaluated for feasibility and acceptability, and manualized. Three phases of research are proposed. In Phase 1, the investigators will conduct formative research to integrate YM-AIM and YIM and refine our assessment battery (Aim 1). In Phase 2, the investigators will finalize the study protocols and consents and develop a manual of operations (Aim 2). In Phase 3, investigators will pilot test Y2Prevent with 30 participants. Assessment measures will also be pilot tested during three assessment sessions, at baseline (first study visit) and 3- and 6-month follow-up (after post-intervention test). Intervention outcomes include drug use in past 30 days and 3 months, alcohol use, condomless sex, number of partners, condom use intention, condom use self-efficacy, HIV testing recency/frequency, and linkage to care. Findings from this pilot research will inform selection of measures and outcomes for a future randomized clinical trial (RCT) and provide estimates of possible intervention effect sizes (group means, SDs) for trial planning. Process measures include data on sources of recruitment and recruitment rates, trial retention rates, and identification of barriers and facilitators to recruitment and retention.

WORKING GROUPS - PHASE 1:

During Phase 1, the investigators will convene two working groups of AAYMS to engage in a process of integrating the Young Men's Adult Identity Mentoring (YM-AIM) and Youth Initiated Mentoring (YIM). Each work group will include 8-10 young men. These men will be recruited from our existing HYM cohort.

Prior experience has taught us that creating groups with shared key characteristics (e.g. risk profile, sexual identity or age) is the most effective means of facilitating more in-depth discussions. Each group, consisting of 6-8 members, will be convened on a weekly basis and each meeting will focus on one specific topic (i.e.,common challenges that AAYMSM experience with HIV prevention; what AAYMSM want from a mentor) - there will be around 7 weekly lessons that participants will attend. During these meetings, participants will review each unit of the original YM-AIM and YIM curricula and discuss what components would be most relevant. Groups will be facilitated by the research assistant, and each week a volunteer from each group will be asked to serve as a co-facilitator in an effort to increase ownership for intervention adaptation and to assist in maintaining order within the group.

Guided discussions will focus on different aspects of the curricula such as: 1) common challenges that AAYMSM experience with HIV prevention; 2) what AAYMSM want from a mentor; 3) managing positive and negative influences in their lives; 4) challenges in accessing care; and 5) the role that intimate partners play in their lives. The investigators will brainstorm potential activities that can be integrated into our newly adapted Y2Prevent curriculum that focus on these areas (e.g., PrEP Myth or Truth game).

PILOT TEST - PHASE 3: In Phase 3, the investigators will pilot test Y2Prevent with three working groups of African American young men who have sex with men (AAYMSM) in Los Angeles. Each group will have up to 10 members (n=30). The intervention will be delivered to the three groups in a sequential order so that the experiences from the first group can be used to adapt and/or further refine the intervention before it is pilot tested with the second group. Feedback from the first group will be used to further adapt and refine the intervention. It will be pilot tested again with a second group of 10 participants. Y2Prevent will be further refined as needed, and it will then be pilot tested with a third and final group of up to ten participants. The investigators will continue to gather information, solicit input, and refine Y2Prevent until the investigators are satisfied that the intervention is truly relevant, acceptable, and appropriate for the target population. These group discussions will be audio-recorded and professionally transcribed for analysis. The focus groups are expected to last 1.5 - 2 hours each.

ELIGIBILITY:
Inclusion Criteria:

* 18-24 years old;
* identify as a cisgender male;
* identify as Black/African American;
* identify as gay, bisexual, or some other same-sex identity, and/or report having had sex with a man;
* HIV-negative;
* not currently enrolled in an HIV prevention study;
* living in the Los Angeles metro area;
* has access to a device (laptop, tablet or phone) with internet access in order to participate in virtual group sessions, complete online surveys, and receive payment via Venmo or Cash App; and
* has access to a telephone in order to be able to participate in and complete the qualitative exit interview, which will be conducted via telephone.

Exclusion Criteria:

* outside age 18-24 years old;
* identify as a transgender man or woman;
* identify as White/Caucasian, Latino/Hispanic, Asian/Pacific Islander, Native American, Indigenous, or any other ethnicity besides African American;
* identify as straight;
* HIV-positive;
* currently enrolled in an HIV prevention study;
* currently living outside the Los Angeles metro area;
* does not have access to a device (laptop, tablet or phone) with internet access, which is necessary to participate in weekly group sessions, complete online surveys and receive payment for participation via Venmo or Cash App; and
* does not have access to a telephone, which is necessary to participate in the qualitative exit interview at the end of the seventh and final study session.

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We are recruiting only African American men ages 18-24 for this study. This study includes only men who have sex with men as participants due to their potential risk for HIV and the disproportionately high rates of HIV among African American men. Young men, ages 18-24, will be the target age due to the lack of data on this particular population of men.
Enrollment: 27 (Actual)
Dates: Start 2020-01-22 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Sexual risk behaviors | Baseline
  Condomless anal intercourse; frequency of this behavior during reporting period; # of sexual partners during the reporting period; use of PrEP/PEP during reporting period
Alcohol and illincit drug use | Baseline; will asses past 30-day use; past 3 month
  Frequency of acohol and illiict drug use including cocain, ecstasy, methamphetamines, psychedilic drugs (e.g., LSD, shrooms); heroin, opiates, prescription drugs without a prescription; marijuana
Sexual risk behaviors | 3 months post intervention
  Condomless anal intercourse; frequency of this behavior during reporting period; # of sexual partners during the reporting period; use of PrEP/PEP during reporting period
Alcohol and illincit drug use | 3 months post intervention
  Frequency of acohol and illiict drug use including cocain, ecstasy, methamphetamines, psychedilic drugs (e.g., LSD, shrooms); heroin, opiates, prescription drugs without a prescription; marijuana
Sexual risk behaviors | 6 months post intervention
  Condomless anal intercourse; frequency of this behavior during reporting period; # of sexual partners during the reporting period; use of PrEP/PEP during reporting period
Alcohol and illincit drug use | 6 months post intervention
  Frequency of acohol and illiict drug use including cocain, ecstasy, methamphetamines, psychedilic drugs (e.g., LSD, shrooms); heroin, opiates, prescription drugs without a prescription; marijuana
Illincit drug use | urine analysis for recent drug use (up to 1 week) at time of assessment (baseline)
  Presence of marijuana, methamphetamines, cocaine, heroin, opiates, barbituates, benzodiazepines, ecstasty, GHB, PCP
Illincit drug use | urine analysis for recent drug use (up to 1 week) at time of assessment (3 months post intervention)
  Presence of marijuana, methamphetamines, cocaine, heroin, opiates, barbituates, benzodiazepines, ecstasty, GHB, PCP
Illincit drug use | urine analysis for recent drug use (up to 1 week) at time of assessment (6 months post intervention)
  Presence of marijuana, methamphetamines, cocaine, heroin, opiates, barbituates, benzodiazepines, ecstasty, GHB, PCP

SECONDARY OUTCOMES:
PrEP Uptake | Current PrEP use at time of assessment (3 months post)
  Measured with urine analysis
PrEP Uptake | Current PrEP use at time of assessment (6 months post)
  Measured with urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Michele D Kipke, PhD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Researchers interested in the Y2Prevent data can request access to baseline and follow up survey data, specimen collection data and qualitative data from the intervention pilot groups in the form of written transcriptions. A publication plan and data use agreement would be reviewed and approved by the PI prior to sharing any data.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: 7/1/23-6/30/26
Access Criteria: Email requests can be submitted to the Senior Programs Manager Lindsay Slay at lslay@chla.usc.edu or PI Michele Kipke at mkipke@chla.usc.edu. Templates will be provided for the publication plan and data use agreement.